CLINICAL TRIAL: NCT04831918
Title: A Prospective Clinical Study Evaluating Clinical, Radiographic And Patient-Reported Outcomes Of THA With Cemented Acetabular Cups
Brief Title: Cemented Acetabular Cups Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Total Hip Arthroplasty
Keywords: Cemented acetabular cup

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mueller cemented cups (Experimental): Patients undergo total hip arthroplasty with the implant of the Mueller cemented cup as acetabular component.
  Interventions: Device: Mueller cemented cups

INTERVENTIONS:
Device: Mueller cemented cups — Patients undergo total hip arthroplasty with the implant of Mueller cemented cups

SUMMARY:
This clinical study has the aim to evaluate clinical, radiographic, patient-reported outcomes of total hip arthroplasty with the implant of Mueller cemented acetabular cups up to 2 years after surgery, in order to assess the performance of the device. Furthermore, it aims to collect short-term survivorship of the implant and the incidence of early complications.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has participated in the Informed Consent process and has signed the Informed Consent form previously approved by the Ethics Committee;
2. The patient diagnosis is one or more of the following:

   * Patient with advanced articular destruction generated by primary degenerative or post-traumatic arthrosis or rheumatoid arthritis;
   * Patient with avascular necrosis of the femoral head or fracture of the femoral neck;
   * Patient with congenital or acquired deformity;
   * Patient with failures of previous operations, like osteosynthesis, articular reconstruction, arthrodesis, hemi-arthroplasty or total arthroplasty.
3. The patient is willing and able to complete scheduled follow-up evaluations as described in the Patient Information Sheet;

Exclusion Criteria:

The patient should be excluded from the study if he/she meets any of the following criteria, which reflect the cemented acetabular cup contraindication for use:

1. Acute or chronic infections, local or systemic infections;
2. Serious muscular, neurological or vascular diseases affecting the concerned limb;
3. Any concomitant disease and dependence that might affect the implanted prosthesis;
4. Allergy to material;
5. Metal-on-metal systems: patients with renal impairment.
6. Patient's age<18
7. Female patients who are pregnant, nursing, or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical progression of Harris Hip Score (HHS) from baseline to 2 years after surgery | 2 years Follow up
  HHS ranges from 0 to 100, being 0 the worst and 100 the best conditions. HHS is reported as 90-100 for excellent results, 80-90 for good, 70-79 for fair, 60-69 for poor, and below 60 for a failed result. The outcome is considered satisfactory for values over 80

SECONDARY OUTCOMES:
Radiographic evaluation and stability assessment of the implant up to 2 years FU | 6 weeks, 1 year and 2 years FU
  Radiographic stability, radiographically detectable complications
Clinical progression of HOOS up to 2 years FU, compared to the baseline | 6 weeks, 1 year and 2 years FU
  Hip disability and osteoarthritis outcome score (HOOS) is a patient-reported outcome measurement, that ranges from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms
Change in TUG from preoperative up to 2 years FU | 6 weeks, 1 year and 2 years FU
  Timed Up and Go
Clinical progression of HHS up to 1 year FU, compared to the baseline | 6 weeks, 1 year
  Harris Hip Score
Implant survivorship (Kaplan-Meier estimate) at 2 years after surgery | 2 years FU
Incidence of device-related AE/SAE up to 2 years of follow-up | 6 weeks, 1 year and 2 years FU
  Adverse events and device deficiencies

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marega, Principal Investigator — Ospedale San Camillo di Trento
Locations (1):
- Ospedale San Camillo di Trento, Trento, TN, Italy

IPD SHARING:
Plan to Share IPD: No